CLINICAL TRIAL: NCT03150706
Title: A Phase II Study of Avelumab in Patients With Mismatch Repair Deficient or POLE Mutated Metastatic Colorectal Cancer
Brief Title: Avelumab for MSI-H or POLE Mutated Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mCRC avelumab
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: POLE mutation; mismatch repair deficient; Avelumab
MeSH Terms: conditions — Colorectal Neoplasms; Turcot syndrome | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): The mismatch repair deficient or microsatellite instable, or POLE mutated metastatic colorectal cancer patients who were progressed after at least one prior systemic treatment for metastatic setting.
  After checking the eligibility for the study entry, patients will be entered into the study treatment with avelumab monotherapy.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Patients will receive 10 mg/kg of avelumab via intravenous infusion every 2 weeks.
  Response evaluation will be performed every 6 weeks (± 1-week window period). Treatment will be continued until disease progression, unacceptable adverse events or the patient's refusal.
  Treatment through progression is at the investigator's discretion, and the investigator should ensure that patients do not have any significant, unacceptable, or irreversible toxicity that indicate that continuing treatment will not further benefit the patient. The Investigator should ensure that patients still meet all of the inclusion criteria and none of the exclusion criteria for this study.
  Other Names: MSB0010718C

SUMMARY:
The POLE mutations represent high somatic mutation loads in patients with colorectal cancer, especially in those with MMR proficient or MSS, therefore, tumors harbouring POLE mutations might be susceptible to immune checkpoint blockade.

Based on these reasons, Investigator planned a phase II study of avelumab monotherapy in patients with previously treated, metastatic, MMR deficient (MSI-H) or POLE mutated colorectal cancer.

DETAILED DESCRIPTION:
Later-line therapies after failure of standard treatments for metastatic colorectal cancer patients are limited; regorafenib and TAS-102 have shown clinical activity for these patients, however, efficacy outcomes seemed not to be sufficient although there have been rather higher frequencies of adverse events.

Mismatch repair (MMR) deficiency or microsatellite instability-high (MSI-H) played a role of negative predictive factor for adjuvant fluorouracil-based chemotherapy in patients with resected colorectal cancer. In the metastatic setting, deficient MMR or MSI-H represented poor prognosis; however, their predictive role has been documented after the pembrolizumab trial was reported. The results of the pembrolizumab trial demonstrated that the PD-1 blockade with pembrolizumab monotherapy showed 40% of confirmed immune-related objective response rates in patients with MMR deficient metastatic colorectal cancers; hence there was no objective response in those with MMR proficient tumors. The progression-free rates at 20 weeks were 78% versus 11%, respectively, also favouring those with MMR deficient tumors. However, the MMR deficiency of MSI-H is found in only about 5% in patients with metastatic colorectal cancer, which is too small to expand potential candidate of immunotherapy.

One of the proposed mechanism of promising efficacy from pembrolizumab for MMR deficient colorectal cancer is that MMR deficient or MSI-H colorectal cancers harbour higher somatic mutation loads than MMR proficient colorectal cancer (a mean of 1782 somatic mutations per tumor in the MMR deficient tumors versus 73 in the MMR proficient tumors in the results of pembrolizumab trial); somatic mutations have the potential to encode non-self immunogenic antigens; therefore, immunotherapy enhancing immune surveillance produced promising treatment efficacy in the MMR deficient tumors.

The POLE gene encodes the catalytic subunit of DNA polymerase epsilon, and it involves DNA repair and chromosomal replication. The POLE mutations are located in the exonuclease domain, and their presence has already been reported in the various cancers including colorectal and endometrial cancer.

The POLE mutations represent high somatic mutation loads in patients with colorectal cancer, especially in those with MMR proficient or MSS, therefore, tumors harbouring POLE mutations might be susceptible to immune checkpoint blockade.

Based on these reasons, Investigator planned a phase II study of avelumab monotherapy in patients with previously treated, metastatic, MMR deficient (MSI-H) or POLE mutated colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the colon or the rectum.
2. Mismatch repair deficient or microsatellite instable (defined below), or POLE mutated tumors A. Mismatch repair deficient: loss of expression by immunohistochemical stains 4. ≥ 1 out of 4 markers (MLH1, MSH2, MSH6, PMS2) B. Microsatellite instable: loss of stability ≥2 out of 5 gene panels (BAT-25, BAT-26, D2S123, D5S345, D17S250)
3. Progressed after at least first-line systemic chemotherapy for metastatic setting.
4. ≥ 1 measurable lesion(s) by RECIST 1.1.
5. Unresectable advanced or metastatic disease.
6. Age over 20 years old.
7. ECOG 0-1, but final decision by clinical.
8. Adequate organ functions. A. Bone marrow function: Hemoglobin 9.0 g/dL, ANC 1,500/mm3, platelet 100,000/mm3 B. Hepatic functions: bilirubin ≤ 1.5 X ULN, AST/ALT ≤ 2.5 X ULN (≤ 5 X ULN in cases of liver metastasis) C. Renal functions: serum Cr ≤ 1.5 X ULN or calculated CCr (Cockroft) ≥ 30 ml/min
9. Be willing and able to comply with the protocol for the duration of the study.
10. Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw the study at any time, without prejudice.
11. Female subjects must either be of non-reproductive potential ( 60 years old and no menses for 1 year without an alternative medical cause, or history of hysterectomy, or history of bilateral tubal ligation, or history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
12. Women of childbearing potential and men must agree to use highly efficient contraception since signing of the IC form until at least 8 weeks after the last study drug administration.

Exclusion Criteria:

1. Any prior treatment with PD-1 or PD-L1 inhibitor.
2. Receipt of the last dose of chemotherapy ≤ 28 days prior to the first dose of study drugs.
3. Current or prior use of immunosuppressive medication within 28 days before the first dose of avelumab, with the exceptions for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
4. Concurrent or previous history of another primary cancer within 3 years prior to randomisation except for curatively treated cervical cancer in situ, non-melanomatous skin cancer, superficial bladder cancer (pTis and pT1) and curatively treated thyroid cancer of any stage. Concurrent, histologically confirmed, unresected thyroid cancer without distant metastasis could be allowed with the agreement of the chief principal investigator.
5. Uncontrolled CNS metastases; permitted if asymptomatic or neurologically stable.
6. Prior radiation therapy would be permitted, but non-radiated evaluable lesions should be present at study entry.
7. Radiation therapy during study treatment is not permitted, but if the local investigator decides that radiation therapy should be given during study treatments, he should be convinced that there is no evidence of disease progression with agreement of the chief principal investigator.
8. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
9. Active or prior documented autoimmune disease within the past 2 years; subjects with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
10. Active or prior documented inflammatory bowel disease.
11. History of prior immunodeficiency.
12. History of allogeneic organ transplantation.
13. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
14. History of previous clinical diagnosis of active tuberculosis.
15. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines
16. Known history of testing positive for HIV
17. Hepatitis B virus (HBV) or hepatitis C virus(HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)Except, resolved HBV infection (as evidenced by detectable HBV surface antibody, detectable HBV core antibody, undetectable HBV DNA, and undetectable HBV surface antigen) or Chronic HBV infection (as evidenced by detectable HBV surface antigen or HBV DNA). Subjects with chronic HBV infection must have HBV DNA < 100 IU/mL and must be on antiviral therapy.
18. Major surgery or significant traumatic injury within 28 days prior to study treatment.
19. Non-healing wound, ulcer, or bone fracture.
20. Current evidence of significant gastrointestinal bleeding or (impending) obstruction.
21. Concomitant participation in another clinical trial.
22. Pregnant of breast-feeding subjects. Women of child-bearing potential must have pregnancy test within 7 days and a negative result must be documented before start of study treatment.
23. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
24. Active infection requiring systemic therapy.
25. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
26. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum CEA, TSH, T3, free T4, EKG,CT (or MRI) scans of evaluable/measurable lesions by RECIST 1.1. | 6 weeks(maximum 7 weeks)
  During the CRT

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No